CLINICAL TRIAL: NCT06569940
Title: Single-center Evaluation of Sleepiz One+ Algorithm in Estimating Respiration Rate and Heart Rate Compared to Gold Standard
Brief Title: Sleepiz One+ vs. Capnography and Electrocardiography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sleepiz AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-001-CI
Record Dates: First submitted 2024-08-13; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Sleep Apnea; Asthma; COPD; Hypertension; Diabetes; Respiratory Disease; Cardiovascular Diseases
MeSH Terms: conditions — Sleep Apnea Syndromes; Asthma; Pulmonary Disease, Chronic Obstructive; Hypertension; Diabetes Mellitus; Respiration Disorders; Cardiovascular Diseases

STUDY DESIGN:
Masking Description: Annotators of capnography data were blinded to the values provided by the investigational device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleepiz One+ vs. gold standard (Other): Each enrolled participant will undergo a simultaneous recording with the Sleepiz One+, Capnography device and cardiorespiratory polygraphy to measure respiration rate at and heart rate at rest, while sitting and lying down on a bed.
  Interventions: Device: Sleepiz One+

INTERVENTIONS:
Device: Sleepiz One+ — In this study Sleepiz One+ will measure heart rate and respiration rate of a participant sitting or lying in different positions (right and left side, back, abdomen) on a bed. The recording will take around 42 minutes.

SUMMARY:
Respiratory Rate (RR) and heart rate (HR) are vital signs crucial for assessing a patient's overall health, providing insights into various conditions and stressors. Effective management of chronic diseases relies on detecting pathological changes early, with RR being among the most sensitive predictors of patient deterioration. Therefore, vigilant monitoring of RR and HR is vital for improving patient outcomes.

The primary aim of this study is to provide a thorough comparison of the performance of Sleepiz One+ algorithms and end-tidal carbon dioxide measurement (EtCO2) Capnography for measuring respiration rate and electrocardiography (ECG) for measuring heart rate, in healthy adults and patients suffering from chronic conditions (e.g., hypertension, Chronic Obstructive Pulmonary Disease (COPD), asthma, diabetes), at rest in a clinical setting when the data is acquired with the new hardware version. Additionally, the investigators will evaluate the performance of RR estimation against the thoracic effort belt and the HR against the pulse oximetry.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Age >=18years
* Informed Consent as documented by signature
* One (or more) chronic medical condition/s (e.g., diabetes, asthma, cardiovascular or respiratory diseases, etc.)

Healthy volunteers

* Age >=18years
* Informed Consent as documented by signature
* No diagnosed chronic medical condition

Exclusion Criteria:

Patients

* Previous enrolment into the current study,
* Cardiac pacemaker or another implanted electrical device
* Women who are pregnant or breastfeeding
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, delirium etc. of the participant

Healthy volunteers:

* Previous enrolment into the current study,
* Cardiac pacemaker or another implanted electrical device
* Women who are pregnant or breastfeeding
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, delirium etc. of the participant
* Presence of diagnosed chronic medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Instantaneous respiration rate measurement accuracy per 60s epoch | During 60 seconds
  Instantaneous respiration rate measurement accuracy per 60s epoch against visually scored capnography data, recorded on subjects lying down and resting on a bed
Instantaneous heart rate measurement accuracy per 60s epoch | During 60 seconds
  Instantaneous heart rate measurement accuracy per 60s epoch against ECG R-R interval, recorded on subjects lying down and resting on a bed

CONTACTS AND LOCATIONS:
Overall Officials: Christian Neumann, Dr. med., Principal Investigator — Zentrum für Schlafmedizin "Schlaflabor Fluntern"
Locations (1):
- Schlaflabor Fluntern, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No